CLINICAL TRIAL: NCT02909283
Title: Determinants of Cerebral Oxygenation and Perfusion in SCA Children Based on Combined ASL MRI, NIRS and Hemorheological Investigation
Brief Title: Sickle Cell Anemia and Cerebral Microcirculation : Multimodal Exploration
Acronym: DREAM²
Status: Completed | Type: Observational
Sponsor: Imagine Institute (Other)
Collaborators: Hopital Universitaire Robert-Debre (Other)
Responsible Party: Sponsor
Other Study IDs: IMIS2014-04
Record Dates: First submitted 2016-09-05; First posted 2016-09-21 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are taken, in order to create Biobank (DNA, serum and plasma)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sickle cell disease patients: Physical exams and blood analyzes
  Interventions: Procedure: Physical exams and blood analyzes

INTERVENTIONS:
Procedure: Physical exams and blood analyzes — Blood samples collection (for DNA, plasma and cells analyzes) ; Hemorheologic analyzes ; ASL sequence on MRI ; Near Infra Red Spectroscopy (NIRS) and associated cardiofrequency analyze.

SUMMARY:
The aim of this study is to evaluate determinants of cerebral oxygenation and perfusion at the microcirculatory level in children with sickle cell anemia (SCA) using combined novel investigational tools: Arterial Spin Labeling (ASL) perfusion MR (Magnetic Resonnance) imaging, brain Near Infra-Red Spectroscopy (NIRS) and red blood cell (RBC) rheological properties.

DETAILED DESCRIPTION:
The investigators hypothesize that brain perfusion and/or oxygenation modifications may be evidenced in SCA children who have no microarteriopathy and may correlate with hemorheological abnormalities and impaired vasomotion. A multimodal approach designed to study a. cerebral perfusion and oxygenation, b. flow motion properties and c. blood rheological parameters might help to describe the different processes involved in cerebral ischemia.

ELIGIBILITY:
Inclusion Criteria:

* SS or S-beta° genotype;
* age 6-16 years;
* steady state;
* normal TCD (Transcranial Doppler);
* parental study approval and written informed consent.

Exclusion Criteria:

* SC, Sbeta+, SD Punjab genotype
* history of overt stroke,
* intracranial or cervical arterial stenosis,
* abnormal TCD at the time of the study.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient included will be patients suffering from Sickle Cell Anemia, and coming at the study center in the frame of their annual follow-up visit.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
Number of patients on which we detect default of cerebral perfusion (in order to correlate them with other clinical or biological parameters) | 1.5 years
  ASL sequence (duration 4 min) : Regional brain tissue perfusion (expressed in mL/min/100g of tissue) will be measured in different lobes in both hemispheres and in the cerebellum. Pattern of perfusion will be analysed and measured.

SECONDARY OUTCOMES:
Bifrontal cerebral hemoglobin oxygen saturation | 1.5 years
  Bifrontal cerebral hemoglobin oxygen saturation monitored by NIRS (15 min). Spectral analyses (Fourrier transform) will be used to analyze the brain microvascular oxygen variability and calculate the flowmotion and vasomotion activities.
Description of the global assessment of RBC deformability | 1.5 years
  The description of the global assessment of RBC deformability will be done via a global association of several biological parameters : RBC deformability at several shear stresses by ektacytometry, RBC aggregation properties by syllectometry and blood viscosity by cone-plate viscosimetry. Measurements will be made according to the international guidelines for standardisation in hemorheology and within 4/5 hrs of sampling

CONTACTS AND LOCATIONS:
Overall Officials: Valentine Boursse, Principal Investigator — Hôpital Necker-Enfants Malades; Suzanne Verlhac, Study Director — Centre Hospitalier intercommunal de Créteil
Locations (2):
- France (2):
  - Centre Hospitalier Intercommunal, Créteil
  - Necker - Enfants Malades hospital, Paris

IPD SHARING:
Plan to Share IPD: No